CLINICAL TRIAL: NCT03910543
Title: Open-label Trial of Tofacitinib in Cutaneous Sarcoidosis and Granuloma Annulare
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2000023910
Record Dates: First submitted 2019-04-04; First posted 2019-04-10 (Actual); Last update posted 2021-07-14 (Actual); Status verified 2021-07

CONDITIONS: Cutaneous Sarcoidosis; Granuloma Annulare
MeSH Terms: conditions — Granuloma Annulare | interventions — tofacitinib

STUDY DESIGN:
Intervention Model Description: open-label trial
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Patients with Cutaneous Sarcoidosis (Experimental): Patients with cutaneous sarcoidosis that may also have also have internal organ sarcoidosis
  Interventions: Drug: Tofacitinib 5 mg twice daily
- Patients with Granuloma Annulare (Experimental): Patients with granuloma annulare that is long-standing and/or widespread
  Interventions: Drug: Tofacitinib 5 mg twice daily

INTERVENTIONS:
Drug: Tofacitinib 5 mg twice daily — Tofacitinib will be administered at a dose of 5 mg twice daily
  Other Names: Xeljanz 5 mg twice daily

SUMMARY:
To investigate the ability of tofacitinib, a Janus kinase (JAK) inhibitor, to treat patients with cutaneous sarcoidosis and granuloma annulare during 6 months of therapy.

DETAILED DESCRIPTION:
An open-label clinical trial of tofacitinib in cutaneous sarcoidosis and GA. The hypothesis is that Janus Kinase (JAK) 1/3 inhibition with tofacitinib will be effective for the treatment these two diseases. Tofacitinib will be administered at a dose of 5 mg twice daily and response to therapy will be assessed at months 1, 3, and 6 of therapy. The primary outcomes will be improvement in the Cutaneous Sarcoidosis Activity and Morphology Instrument (CSAMI) and Granuloma Activity Scoring Index (GASI) after 6 months of tofacitinib therapy. Secondary outcomes will include improvement in internal organ sarcoidosis (i.e. lung, cardiac) and skin related quality of life. Pre- and on treatment PET-CT scans will be performed in patients with sarcoidosis with internal organ involvement. Pre- and on treatment blood collection and skin biopsies will be performed for correlative scientific studies using RNA sequencing, immunohistochemistry (IHC), and cytokine profiling.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old or older
* Diagnosis of cutaneous sarcoidosis or granuloma annulare with supportive skin biopsies in which other causes of granulomas (infectious, foreign body) have been ruled out
* Patients with either: Cutaneous Sarcoidosis Activity and Morphology (CSAMI) activity score greater than or equal to 10 (patients with a CSAMI greater than or equal to 10 have active cutaneous sarcoidosis involving several distinct cutaneous sites and would otherwise be considered candidates for systemic therapy), or any CSAMI score and sarcoidosis involvement causing functional impairment (i.e. nasal or visual field obstruction).
* For patients with granuloma annulare, patients with 5% or greater Body Surface Area (BSA) will be enrolled.
* If patients are on other systemic therapies for their sarcoidosis or granuloma annulare, they must be taking a stable dose of the other medication(s) for at least 3 months with no plans to change the regimen in the next 6 months. With the exception of methotrexate and/or low dose prednisone, use of concomitant immunosuppressants, e.g. infliximab, azathioprine, etc., will not be permitted.
* Females of childbearing potential must agree to use birth control during the study and there must be a negative pregnancy test documented prior to starting the medication.
* Patients must be willing to undergo skin biopsies, blood collection, and total body photography and comply with clinic visits

Exclusion Criteria:

* Age <18 years old
* Patients with a history of malignancy (except history of successfully treated basal cell or squamous cell carcinoma of the skin)
* Patients known to be HIV or hepatitis B (HBV) or C (HCV) positive (prior exposure to but clearance of HBV and HCV is acceptable for study entry as long as patient is being monitored by hepatology)
* Patients with active tuberculosis or untreated latent tuberculosis as determined by positive tuberculin skin test or positive QuantiFERON® Tuberculosis (TB) test and, as necessary, chest X-ray
* Patients with significant hepatic impairment
* Patients with untreated peptic ulcer disease
* Patients taking immunosuppressive medications, with the exception of methotrexate and/or low- dose prednisone, including but not limited to mycophenolate mofetil, azathioprine, tacrolimus, cyclosporine, or Tumor Necrosis Factor (TNF-α) inhibitors
* Women of childbearing potential who are unable or unwilling to use birth control while taking the medication
* Women who are pregnant or nursing. If a woman becomes pregnant during the study, she will stop study medication and be removed from the study. She will be urged to follow up with her Primary Care Physician or OB/GYN. The study doctors will ask to follow the pregnancy to its outcome.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2019-04-11 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
Change in Cutaneous Sarcoidosis Activity and Morphology Instrument (CSAMI) | 6 - 12 months
  For patients with sarcoidosis: change in CSAMI score after 6 months of treatment with tofacitinib compared to baseline.
  The activity portion of the CSAMI score will be utilized. The range of scores is from 0 to 165. Higher scores correspond with higher cutaneous disease burden.
  The percentage change in CSAMI score will be calculated as follows:
  change in CSAMI score = [baseline CSAMI - final CSAMI] / baseline CSAMI
  Higher percentage change corresponds to more improvement on therapy (0% = no change, 100% = complete disease resolution) Negative percentage change corresponds to disease worsening (-25% = 25% worsening of disease)
Percent Change in Body Surface Area (BSA) involvement by GA lesions | 6 - 12 months
  For patients with GA: change in BSA involvement after 6 months of treatment with tofacitinib compared to baseline.
  The range of BSA involvement for this study is from 5% to 100%. Higher BSA involvement corresponds with higher cutaneous disease burden.
  The percentage change in BSA will be calculated as follows:
  Change in BSA = [baseline BSA- final BSA] / baseline BSA Higher percentage change corresponds to more improvement on therapy (0% = no change, 100% = complete disease resolution) Negative percentage change corresponds to disease worsening (-25% = 25% worsening of disease).

SECONDARY OUTCOMES:
Change in Skindex-16: a skin-related quality of life metric | 6 - 12 months
  For all patients: change in Skindex-16 score after 6 months of treatment with tofacitinib compared to baseline
Change in Histologic Findings | 6 -12 months
  Skin biopsies of lesional skin will be performed at baseline and again after 6 months of treatment. Standard hematoxylin and eosin (H&E) and immunohistochemistry for CD68, phospho-STAT1, and phospho-STAT3 will be performed.
Change in RNA sequencing markers (gene expression analysis) | 6 - 12 months
  RNA sequencing will be performed on RNA extracted from skin biopsies of lesional skin at baseline and again after 6 months of treatment.
Change in cytokine biomarkers | 6 - 12 months
  Luminex-based cytokine analysis using a commercially available service will be performed on plasma collected at baseline and again after 6 months of treatment.
Change in activity of internal organ sarcoidosis | 6 - 12 months
  For patients with sarcoidosis: change in PET-CT imaging after 6 months of treatment with tofacitinib compared to baseline

CONTACTS AND LOCATIONS:
Overall Officials: William Damsky, MD, PhD, Principal Investigator — Yale University
Locations (1):
- Yale Center for Clinical Investigation, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Damsky W, Thakral D, Emeagwali N, Galan A, King B. Tofacitinib Treatment and Molecular Analysis of Cutaneous Sarcoidosis. N Engl J Med. 2018 Dec 27;379(26):2540-2546. doi: 10.1056/NEJMoa1805958. PMID 30586518
- [Derived] Damsky W, Wang A, Kim DJ, Young BD, Singh K, Murphy MJ, Daccache J, Clark A, Ayasun R, Ryu C, McGeary MK, Odell ID, Fazzone-Chettiar R, Pucar D, Homer R, Gulati M, Miller EJ, Bosenberg M, Flavell RA, King B. Inhibition of type 1 immunity with tofacitinib is associated with marked improvement in longstanding sarcoidosis. Nat Commun. 2022 Jun 6;13(1):3140. doi: 10.1038/s41467-022-30615-x. PMID 35668129
- [Derived] Wang A, Rahman NT, McGeary MK, Murphy M, McHenry A, Peterson D, Bosenberg M, Flavell RA, King B, Damsky W. Treatment of granuloma annulare and suppression of proinflammatory cytokine activity with tofacitinib. J Allergy Clin Immunol. 2021 May;147(5):1795-1809. doi: 10.1016/j.jaci.2020.10.012. Epub 2020 Dec 11. PMID 33317858